CLINICAL TRIAL: NCT04299997
Title: Accuracy of the PI-RADS v2.1 Score for Characterizing ISUP ≥2 Prostate Cancers on Multiparametric MRI: a Multiple Reader Study
Brief Title: Evaluation of the PI-RADS v2.1 Score Using Multiple Readers
Acronym: MULTI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: MULTI_2020
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer; Urological Cancer
Keywords: multiparametric MRI; ISUP; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 171 mpMRIs corresponding to consecutive patients who underwent: The mpMRIs were performed on a 1.5T GE MR unit or on a 3T GE or Philips MR units. All mpMRIs included T2-weighted imaging, diffusion-weighted imaging (maximal b value: 2000 s/mm²) and dynamic contrast-enhanced imaging.
  Interventions: Other: Assessment of the accuracy of the PI-RADS v2.1 score for predicting the presence of ISUP ≥2 prostate cancer at subsequent biopsy in the dataset of the 171 MRIs for 21 different readers.

INTERVENTIONS:
Other: Assessment of the accuracy of the PI-RADS v2.1 score for predicting the presence of ISUP ≥2 prostate cancer at subsequent biopsy in the dataset of the 171 MRIs for 21 different readers. — 1. Ass of targeted suspect lesions
     On each mpMRI,radiologist will contour lesions that were targeted at subsequent biopsy based on reports. Contours will be disclosed to readers who will assess,for each lesion:
     * Likert score("gut feeling"ie subjective ass of the likelihood that lesion is clinically significant prostate cancer(5-level scale))
     * PI-RADSv2, PI-RADSv2.1 score(by strictly applying the published PI-RADS criteria)
     * EPE score(ie the likelihood of extraprostatic extension;5-level subjective scale without predefined criteria)
     * Max diameter
  2. Def of add suspect lesions Readers could define suspect"additional targets"(AT);for each AT,they will provide the same criteria. It is expected that, for these suspect AT,at least one score is≥3
  3. Ass of lobes Scores of prostate lobes will be automatically calculated based on 2 previous steps of reading. However,in lobes with no suspect lesion,readers could define whether same criteria are1or2,in peripheral zone and transition zone

SUMMARY:
The interpretation of prostate multiparametric MRI (mpMRI) is difficult and requires expertise. As a result, it suffers from substantial inter-reader variability. The so-called Prostate Imaging Reporting and Data System (PI-RADS) scoring system has been launched in 2012 to try and standardise prostate mpMRI interpretation. It is a 5-level score that assesses the likelihood that suspicious focal prostatic lesions seen on mpMRI are clinically significant prostate cancers. Despite the use of semi-objective criteria for each category of the score, the inter-reader reproducibility of the first two versions (PI-RADS v1 launched in 2012 and PI-RADS v2 launched in 2015) was moderate at best, even for experienced readers. The last version (PI-RADS v2.1) has been launched in March 2019 in an effort to improve the inter-reader reproducibility. This version has not been evaluated yet.

The purpose of our study is to evaluate the accuracy and inter-reader reproducibility of the PI-RADS v2.1 score on a large set of 171 prostate MRIs using 21 readers of varying experience.

Twenty-one readers (14 seniors and 7 juniors) from 9 different institutions and with varying experience in prostate mpMRI accepted to participate to the study.

Reader will assess the dataset independently and will be blinded to the other readers' results. They also be blinded to clinical and biochemical data.

ELIGIBILITY:
Inclusion Criteria:

* Prostate mpMRI and biopsy performed at our institution
* Performed between September 2015 and July 2016
* No history of prostate cancer at the time of the mpMRI

Exclusion Criteria:

* Patients who already had treatment for prostate cancer
* Patients under Active Surveillance

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Consecutive patients with mpMRI and subsequent biopsy between September 2015 and July 2016 (see above).
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
AUC of the PI-RADS v2.1 score for predicting ISUP ≥2 cancer at subsequent biopsy at the lesion level. | June 2020.
  Analysis at the lesion level will be favored to get an evaluation of the influence of experience of readers scoring the exact same set of lesions.

SECONDARY OUTCOMES:
AUC of the PI-RADS v2.1 score for predicting ISUP ≥2 cancer at biopsy, at the lesionlobe and patient levels | June 2020
Inter-reader concordance of the PI-RADS v2.1 score, at lesion, lobe and patient levels | June 2020
AUC of the PI-RADS v2 score for predicting ISUP ≥2 cancer at subsequent biopsy at the lesion, lobe and patient levels | June 2020
Inter-reader concordance of the PI-RADS v2 score at lesion, lobe and patient levels | June 2020
AUC of the Likert score for predicting ISUP ≥2 cancer at biopsy at the lesion, lobe and patient levels | June 2020
Inter-reader concordance of the Likert score at lesion, lobe and patient levels | June 2020
Analysis of the diagnostic value of the PI-RADS v2.1 components | June 2020
  The PI-RADS v2.1 score is made by several components who have different diagnostic weights. The added value of the following components will be assessed:
  * Lesions DCE+: do they correspond more often to ISUP ≥2 cancers than DCE- lesions?
  * Lesions with DWI score of 4: is a size of 10-14 mm more predictive of ISUP ≥2 cancers than a size < 10 mm?
  * Lesions with a T2w score of 2 and a DWI score of 4 in the PI-RADS v2.1 score: what is the proportion of ISUP ≥2 cancers?
Added value of the Likert score | June 2020
  - This part will be only exploratory and narrative. It is aimed at evaluating, at least for the most experienced readers, if there are circumstances in which the Likert score (i.e. "gut feeling") is more predictive of ISUP ≥2 cancers than the PI-RADS v2.1 score.
Description of patients with negative initial biopsy and who were diagnosed with ISUP ≥2 cancer after 3 years of follow-up | June 2020
  Because targeted and systematic biopsy may miss cancer foci, follow-up data will be retrieved from the patients' files. Patients with no follow-up data within the last year will be reached by phone to update their follow-up.The patients with initial biopsy showing no cancer or ISUP 1 cancer and who were subsequently diagnosed with ISUP ≥2 cancers during the 3-year follow-up will be reported and described.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France